CLINICAL TRIAL: NCT05228925
Title: GraviD-child Follow-up of the Children´s Health, Growth and Development Within the GraviD-study
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other); Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018-00441
Record Dates: First submitted 2021-11-18; First posted 2022-02-08 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Vitamin D Deficiency; Body Composition; Vascular Health; Cardiometabolic Risk
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Maternal vitamin D status — Maternal vitamin D status (serum 25-hydroxyvitamin D) was collected during the GraviD study, while the woman was pregnant with the child now being followed-up in the GraviD-child study

SUMMARY:
GraviD is a multi-ethnic population-based pregnancy cohort. Pregnant women were invited to participate in the GraviD study when registering for antenatal care in parts of the region of Västra Götaland in Sweden in 2013-2014. All women registering for antenatal care were eligible for inclusion, as long as the pregnancy had not exceeded 16 gestational weeks. In total, 2125 pregnant women were recruited in gestational week 12 during two time-periods; fall 2013 and spring 2014. Blood sampling was performed in gestational week <17 and again at gestational week >31 by midwifes. After delivery, the maternity records were obtained, to collect information on child's gender, birth weight and length and other possible birth outcomes.

DETAILED DESCRIPTION:
In the GraviD-child study, all healthy singleton children born within the GraviD study will be invited to participate in a single clinical follow up. The follow-up will be conducted when all children are between 7-8 years of age. The study centre is located at the Queen Silvia Children´s hospital in Gothenburg, Sweden. The follow up consist of several parts:

1. Measurement of body weight and height, and waist circumference.
2. A questionnaire regarding health, physical activity, sleeping habits and diet.
3. Endothelial function, a measure of how well the blood vessels dilute.
4. Ultra sound of the thickness of the vessels on the neck, wrist and foot
5. Pulse wave velocity, to measure the elasticity of the vessels on the neck and groin.
6. Body composition using bioelectrical impedance.
7. Blood pressure
8. A venous blood sample of maximum 18 ml will be drawn to analyze markers of cardiovascular health. Blood lipids (total cholesterol, triglycerides, HDL cholesterol, LDL cholesterol), lipoprotein A, apolipoproteins (Apo A1 and Apo B), liver enzymes, glucose, insulin, HbA1c, c-reactive protein, leptin, adiponectin, nutritional biomarkers (such as 25-hydroxyvitamin D) will be analyzed.

The study hypothesis is that a low maternal vitamin D status increase the risk of an unfavorable child cardiometabolic risk profile, vascular health and body composition.

Recruitment start in January 2022 and will run for about a year.

ELIGIBILITY:
Inclusion Criteria:

* Born within the GraviD study
* Healthy
* Singleton

Exclusion Criteria:

* Chromosomal abnormality
* Hyper-/Hypothyroidism

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All healthy singleton children born within the GraviD study
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Body composition | At 7-9 years of age
  Fat mass, derived from bioelectrical impedance, will be studied as percentage (%) of the total body weight.
Waist circumference | At 7-9 years of age
  Measurements of waist circumference (in cm) will be assessed.
Blood pressure | At 7-9 years of age
  Blood pressure in mm Hg will be assessed.
Blood lipids | At 7-9 years of age
  Triglycerides in nmol/L will be assessed from a venous blood sample
Blood glucose | At 7-9 years of age
  Glucose in mmol/L will be analyzed from a venous blood sample
Endothelial function | At 7-9 years of age
  Endothelial function will be assessed as reactive hyperemia (RH)-index
Pulse wave velocity | At 7-9 years of age
  Pulse wave velocity (neck to thigh) will be measured in meters per second
Ultrasound | At 7-9 years of age
  Ultra-high frequency ultrasound of dorsalis pedis (in mm) will be measured
Ultrasound | At 7-9 years of age
  Ultra-high frequency ultrasound of radialis (in mm) will be measured
Blood lipids | At 7-9 years of age
  HDL-cholesterol in nmol/L will be assessed from a venous blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Augustin, Ass Prof, Principal Investigator — Göteborg University
Locations (1):
- Queen Silvia Children's Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No